CLINICAL TRIAL: NCT00747383
Title: Influence of Improving Glycaemic Control on Glucagon-Like-Peptide-1 Response to an Oral Glucose Load. Comparison of Sulphonylurea With DPP-4 Inhibition.
Brief Title: How Improvement in Control of Diabetes Influences the Production of a Hormone Produced in the Gut Which Improves the Release and Action of Insulin.
Acronym: MSD-GLP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08/H0201/57
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2008-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; GLP1; DPP4
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — glimepiride; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Glimepiride
- 2 (Active Comparator)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Glimepiride — 3mg oral tablet.
  Other Names: Amaryl.
  Arms: 1
Drug: Sitagliptin — 100mg oral tablet.
  Other Names: Januvia.
  Arms: 2

SUMMARY:
The study is aimed at Type 2 Diabetics who are taking Metformin, but whose Diabetes remains poorly controlled. There are two additional medications already in use, Glimepiride and Sitagliptin will be compared to assess levels of improvement in Diabetes control.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus
* Currently on Metformin but poor glycaemic control,

Exclusion Criteria:

* Under 18 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Comparison of GLP-1 response at baseline and after 3 months treatment of both groups. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, Principal Investigator — Royal Bournemouth Hospital; Joseph Begley, Principal Investigator — Royal Bournemouth Hospital
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom